CLINICAL TRIAL: NCT01677052
Title: THERMOCOOL® SMARTTOUCH™ Catheter for the Treatment of Symptomatic Atrial Fibrillation- Registry
Brief Title: THERMOCOOL® SMARTTOUCH™ Registry
Status: Completed | Type: Observational
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: STR-148
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Symptomatic Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary purpose of this registry is to obtain "real world" clinical use of contact force measurements during ablation procedures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with symptomatic atrial fibrillation (AF) who, in the opinion of the investigator, are candidates for ablation for atrial fibrillation. Candidates who have had previous ablation procedures may be included in the registry
* Subjects who have failed at least one antiarrhythmic drug (AAD)(class I or III, or AV nodal blocking agents such as beta blockers and calcium channel blockers) as evidenced by recurrent symptomatic atrial fibrillation, or intolerable to the AAD.
* Subjects must be 18 years of age or older
* Subjects must be able and willing to comply with all pre-, post and follow-up testing and requirements
* Subjects must provide written informed consent to participate in the registry

Exclusion Criteria:

* Significant congenital anomaly or a medical problem that in the opinion of the investigator would preclude enrollment in this registry
* History of blood clotting or bleeding abnormalities or contraindication to anticoagulation (heparin, warfarin, or dabigatran)
* History of a documented thromboembolic event within the past year
* Significant pulmonary disease (eg, restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease)or any other disease or malfunction of the lungs or respiratory system that produces chronic symptoms
* Previous cardiac surgery (eg, CABG) or valvular cardiac surgical procedure (eg, ventriculotomy, atriotomy, valve repair or replacement, presence of a prosthetic valve)
* Awaiting cardiac transplantation or other cardiac surgery within the next 360 days (12 months)
* Diagnosed atrial myxoma
* Unstable angina
* Uncontrolled heart failure Uncontrolled heart Failure or NYHA Class III or IV heart failure
* Acute illness, active systemic infection, or sepsis
* Any other disease or malfunction that would preclude treatment with ablation in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Target enrollment for this registry is 650 subjects. Of the 650 subjects enrolled, at least 250 will have paroxysmal atrial fibrillation.
Sampling Method: Non-Probability Sample
Enrollment: 426 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Acute Success | 1 year
  Confirmation of entrance block in the pulmonary veins (acute success)
Contact Force | 1 year
  Contact force during ablation procedures
Adverse Events | 1 year
  Procedural complications and adverse events throughout the registry

REFERENCES:
- [Derived] De Potter T, Van Herendael H, Balasubramaniam R, Wright M, Agarwal SC, Sanders P, Khaykin Y, Latcu DG, Maury P, Pani A, Hayes J, Kalman J, Nery P, Duncan E. Safety and long-term effectiveness of paroxysmal atrial fibrillation ablation with a contact force-sensing catheter: real-world experience from a prospective, multicentre observational cohort registry. Europace. 2018 Nov 1;20(FI_3):f410-f418. doi: 10.1093/europace/eux290. PMID 29315382